CLINICAL TRIAL: NCT03152071
Title: Comparison of Robot Assisted Thoracic Surgery With Video Assisted Thoracic Surgery in Case of Lung Cancer: a Prospective Trial With Control Group
Brief Title: Comparison of Robot Assisted Thoracic Surgery With Video Assisted Thoracic Surgery in Case of Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, data nurse, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RATS vs VATS
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Lung Cancer; Postoperative Pain; Blood Loss; Inflammatory Response
Keywords: thoracoscopic surgery; RATS; VATS; Robot
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative; Hemorrhage | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot assisted thoracic surgery (Experimental): RATS
  Interventions: Procedure: Video assited thoracic surgery
- Video assisted thoracic surgery (Active Comparator): VATS
  Interventions: Procedure: Robot assited thoracic surgery

INTERVENTIONS:
Procedure: Robot assited thoracic surgery — The lobectomy will be preformed in case of an operable lung cancer. The thoracic surgery technique used is robot assisted thoracic surgery
  Other Names: RATS
  Arms: Video assisted thoracic surgery
Procedure: Video assited thoracic surgery — The lobectomy will be preformed in case of an operable lung cancer. The thoracic surgery technique used is video assisted thoracic surgery.
  Other Names: VATS
  Arms: Robot assisted thoracic surgery

SUMMARY:
In this study the investigator will compare the effectiveness of robot assisted thoracic surgery (RATS) with video assisted thoracic surgery (VATS) in case of lung cancer.

The perioperative circumstances and postoperative outcome will be compared.

DETAILED DESCRIPTION:
Participants are randomly subdivided (1:1) to either undergo robot assisted lobectomy or video assisted thoracoscopic lobectomy in case of lung cancer. At the end of both surgical interventions the anaesthesiologist administers the same technique of pain relief: paravertebral blockage.

The data that are going to be investigated are: operative time, conversion to spreading of the ribs/thoracotomy, blood loss, lymph node dissection, prolonged air leak, chest tube drainage, length of stay, inflammatory reaction (through inflammatory parameters CRP, IL-3, IL-6, TNF), lung recuperation (through a lung function test) and postoperative pain (VAS score questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years old or older
* Patients can be male or female
* Patients with a lung tumour which is treatable with surgery

Exclusion Criteria:

* Pregnancy
* Inoperable lung tumour
* Patients which are at risk for general anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 2 months
  0 = no pain 10 = unbearable pain: VASscore

SECONDARY OUTCOMES:
blood loss | up to 4 hours
  ml
operative time | up to 4 hours
  duration of surgery
conversion to spreading of the ribs/thoracotomy | up to 4 hours
  0 = no 1 = yes
lymph node dissection | up to 4 hours
  number of lymph nodes
prolonged air leak | up to 7 days
  chest tube present longer than usual
chest tube drainage | up to 7 days
  ml
length of stay | up to 7 days
  duration of hospitalisation after surgery
pulmonary function | 2 months
  recovery of function of the operated lung
Inflammatory reaction | 48 hours
  these inflammatory parameters will be determined: C-reactive protein; IL-3; IL-6; TNF

CONTACTS AND LOCATIONS:
Overall Officials: Wietske Renckens, MD, Study Chair — Universitair Ziekenhuis Brussel; Dirk Smets, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Eef Vanderhelst, MD, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No